CLINICAL TRIAL: NCT02969239
Title: Norepinephrine and Phenylephrine for Cesarean Section
Brief Title: Norepinephrine and Phenylephrine for Maternal Cardiac Output During Spinal Anesthesia for Elective Cesarean Delivery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jeju National University Hospital (Other)
Responsible Party: Principal Investigator, Ae ryoung Lee, Assistant Professor, Jeju National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALee-OB-2016-1
Record Dates: First submitted 2016-10-13; First posted 2016-11-21 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- norepinephrine (Experimental): norepinephrine 5mcg intravenously administered
  Interventions: Drug: Norepinephrine
- phenylephrine (Active Comparator): phenylephrine 100mcg intravenously administered
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Norepinephrine — bolus administered norepinephrine 5mcg intravenously, if SBP <90mmHg or 20% decrease from baseline
  Other Names: vasopressor given
  Arms: norepinephrine
Drug: Phenylephrine — bolus administered phenylephrine 100mcg intravenously, if SBP <90mmHg or 20% decrease from baseline
  Other Names: vasopressor given
  Arms: phenylephrine

SUMMARY:
The purpose of this study is to compare norepinephrine and phenylephrine on the effects of maintaining the cardiac output in Cesarean section under spinal anesthesia.

DETAILED DESCRIPTION:
CO was measured using the NICOM® monitor. Bioreactance, a development from impedance technology, is also emerging as an accessible mode of continuous CO monitoring in the operating room and can provide valuable insight into the hemodynamic effects of our interventions. This method of monitoring provides continuous CO, stroke volume (SV) and heart rate (HR) monitoring, and intermittent BP and SVR assessments at 1-minute intervals.

Either phenylephrine (100 mcg/ml) or norepinephrine (0.5 mcg/ml) in 50-ml syringe that were labeled "study drug". She was not involved in patient's care or study assessment.

The hypotension was defined as systolic blood pressure <80% of baseline or < 90 mmHg, and managed with study drug (1 ml) intravenously. The bradycardia was defined as HR < 60 beats/min and was recorded and managed with atropine (0.5 mg) intravenously as HR < 45 beats/min. The presence of nausea and vomiting was measured on a 3 point scale (1 = no nausea and vomiting, 2 = nausea only, and 3 = both nausea and vomiting) and managed with ondansetron (4mg) intravenously.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I and II, term pregnancy (gestational age>37weeks), planned spinal anesthesia for elective cesarean section

Exclusion Criteria:

* preexisting or gestational hypertension, cerebrovascular or cardiovascular disease, any contraindication to the spinal anesthesia, fetal anormaly, weight<50kg or >100kg, and height<140cm or >180cm.

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
change of cardiac index (L/min/m2) | 1. initial (baseline); 2. 20 min after spinal anesthesia; 3. 1min after the surgery; 4. 1min after baby out; 5. 1min after the end of surgery
  Change from Baseline at time 2, 3, 4, and 5

SECONDARY OUTCOMES:
change of Stroke volume (ml/beat) | 1. initial (baseline); 2. 20 min after spinal anesthesia; 3. 1min after the surgery; 4. 1min after baby out; 5. 1min after the end of surgery
  Change from Baseline at time 2, 3, 4, and 5
change of Total Peripheral Resistance (dynes sec/cm3) | 1. initial (baseline); 2. 20 min after spinal anesthesia; 3. 1min after the surgery; 4. 1min after baby out; 5. 1min after the end of surgery
  Change from Baseline at time 2, 3, 4, and 5
change of Systolic blood pressure (mmHg) | 1. initial (baseline); 2. 20 min after spinal anesthesia; 3. begin the surgery; 4. baby out; 5. the end of surgery
  Change from Baseline at time 2, 3, 4, and 5
change of heart rate (beats per minute) | 1. initial (baseline); 2. 20 min after spinal anesthesia; 3. 1min after the surgery; 4. 1min after baby out; 5. 1min after the end of surgery
  Change from Baseline at time 2, 3, 4, and 5

OTHER OUTCOMES:
Apgar score | 1 min after baby out, 5 min after baby out

CONTACTS AND LOCATIONS:
Overall Officials: AE RYOUNG LEE, Study Director — Jeju National University Hospital
Locations (1):
- Jeju National University Hospital, Jeju City, Jeju-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided